CLINICAL TRIAL: NCT02613130
Title: A Study to Evaluate Oral Malodor and Other Outcomes Following The Use of Two-Step Toothpaste Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015110
Record Dates: First submitted 2015-11-13; First posted 2015-11-24 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Oral Malodor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-Step stannous fluoride toothpaste (Experimental): Two-Step stannous fluoride toothpaste
  Interventions: Drug: Stannous fluoride toothpaste
- Potassium nitrate toothpaste (Active Comparator): Potassium nitrate toothpaste
  Interventions: Drug: Potassium nitrate toothpaste

INTERVENTIONS:
Drug: Stannous fluoride toothpaste
  Arms: Two-Step stannous fluoride toothpaste
Drug: Potassium nitrate toothpaste
  Arms: Potassium nitrate toothpaste

SUMMARY:
This study will assess changes in oral malodor and other factors in response to using a two-step toothpaste oral hygiene relative to a sensitivity whitening toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Have an average hedonic score of at least 6.5;
* Have at least 16 gradable teeth;
* Have at least 10 bleeding sites;
* Have a Lobene composite stain score of ≥1 on at least 1 tooth;
* Have at least one test tooth with recession and a score of 6 or greater on the nine-point comfort/discomfort sensitivity scale;
* Agree to return for scheduled visits and follow the study procedures;
* Agree to refrain from use of any non-study oral hygiene products for the duration of the study;
* Agree to refrain from tongue brushing for the duration of the study;
* Agree to delay any elective dentistry, including dental prophylaxis, until the completion of the study;
* Agree to abstain from eating, drinking, chewing gum, using tobacco products, and any oral hygiene at least eight hours prior to evaluation of oral malodor; and
* Agree to refrain from using deodorant, body lotion/powder/spray, hair products, perfume/cologne, lipstick/gloss, or any other scented products on the mornings of the evaluation days prior to their visit to the clinic.

Exclusion Criteria:

* Oral malodor of systemic origin as determined by health history or examination;
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* Active treatment for periodontitis;
* Removable oral appliances;
* Fixed facial or lingual orthodontic appliances;
* Antibiotic use within four weeks of the Screening visit;
* Any disease or condition that might interfere with the safe participation in the study; and
* Inability to undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Breath odor | Baseline
  Breath measured using a hedonic malodor evaluation
Breath odor | 2 Weeks
  Breath measured using a hedonic malodor evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Resources Group, Whittier, California, United States